CLINICAL TRIAL: NCT02818608
Title: Association Between the Transcranial Direct Current Stimulation (tDCS) and Functional Electrical Stimulation (FES) for Upper-limb Rehabilitation After Stroke - A Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation and Functional Electrical Stimulation for Upper-limb Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APAPS2018
Record Dates: First submitted 2015-11-02; First posted 2016-06-30 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; Cerebrovascular Stroke; Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional electrical stimulation (FES) (Active Comparator): Chronic stroke patients submitted to functional electrical stimulation (FES).
  Interventions: Device: Functional Electrical Stimulation (FES)
- Combination of transcranial direct current stimulation and FES (Experimental): Chronic stroke patients submitted to transcranial direct current stimulation (tDCS) and functional and to functional electrical stimulation (FES).
  Interventions: Device: Combination of Transcranial direct brain stimulation (tDCS) and FES

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) — Functional Electrical Stimulation (FES) + Sham Transcranial direct brain stimulation (tDCS)
  Arms: Functional electrical stimulation (FES)
Device: Combination of Transcranial direct brain stimulation (tDCS) and FES — Real Functional Electrical Stimulation (FES) + Real Transcranial direct brain stimulation (tDCS)
  Arms: Combination of transcranial direct current stimulation and FES

SUMMARY:
The aim of this study is to verify the effectiveness of tDCS combined with FES on upper limb rehabilitation of post-stroke subjects with moderate and severe compromise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ischemic or hemorrhagic stroke diagnosis and moderate or severe hemiparesis (chronic stroke - at least 6 months of disease)
* Ability to reach 60 degrees in the shoulder flexion
* Minimal cognitive ability to understand commands
* No current use of antiepileptic drugs for seizures

Exclusion Criteria:

* Painful shoulder, adhesive capsulitis or glenohumeral subluxation
* Contraindication for electrical stimulation (presence of metallic implants) or risks for the tDCS, as evaluated by means of a standard questionnaire

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Upper-limb reaching analysis evaluated by means of the 3-D motion analysis system (BTS SMART DX 400) | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  3-D motion analysis system

SECONDARY OUTCOMES:
Grip force assessed by means of dynamometer | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  Evaluated by means of dynamometer (Jamar)
Manual dexterity assessed by means of the block and box test | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  Block and box test
Quality of life assessed by means of the Stroke-Specific Quality of Life (SSQOL) | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  Questionnaire
Muscular tone assessed by the Modified Ashworth Scale | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  Modified Ashworth Scale
Assessment of Sensorimotor Recovery After Stroke by the Fugl-Meyer scale | Change from Pre to Post 1 (after the 10th session) and Post 3 (3 months follow-up)
  Fugl-Meyer scale

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Salazar AP, Cimolin V, Schifino GP, Rech KD, Marchese RR, Pagnussat AS. Bi-cephalic transcranial direct current stimulation combined with functional electrical stimulation for upper-limb stroke rehabilitation: A double-blind randomized controlled trial. Ann Phys Rehabil Med. 2020 Jan;63(1):4-11. doi: 10.1016/j.rehab.2019.05.004. Epub 2019 May 31. PMID 31158553